CLINICAL TRIAL: NCT06858566
Title: Impact of the Kaligo Solution on Learning to Write in Children Aged 6 to 11 With Handwriting Disorders: a Multiple Baseline Online SCED Study
Brief Title: Impact of the Kaligo Solution on Learning to Write in Children Aged 6 to 11 With Handwriting Disorders : KALIGO+
Acronym: KALIGO+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ildys (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RI2022_008
Record Dates: First submitted 2025-02-10; First posted 2025-03-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Writing Disorder
Keywords: learning to write; writing disorders; SCED study; Children

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design - SCED
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with handwriting difficulties (Experimental)
  Interventions: Other: Kaligo + score

INTERVENTIONS:
Other: Kaligo + score — The Kaligo + Score will be taken twice a week during baseline and intervention and once a week during follow-up.

SUMMARY:
Writing is a fundamental skill, crucial to a child's success at school and the development of independence. Around 30% of children present difficulties in learning to write, and for some of them (10%), these difficulties persist for a long time. Adapted learning can improve their handwriting. Initial studies into the use of new technologies (tablets, virtual reality headsets) have shown that they can help children learn to write. Attractive to children, these interfaces make it possible to apply new paradigms (e.g. enrichment of feedback [sonification], variation of writing media) that have proved effective, mainly with children with 'typical' development. The Kaligo+ solution is based on the latest scientific advances to offer an innovative approach to learning to write, particularly for children with significant difficulties in this area. This study proposes to test the benefits of the Kaligo+ solution on 15 children with writing difficulties.

The main objective of this pilot study is to demonstrate improved writing performance following use of the Kaligo+ solution in children aged 6 to 11 with writing difficulties, using a Single Case Experimental Design (SCED) methodology.

ELIGIBILITY:
Inclusion Criteria:

* Children with writing difficulties (who may or may not be receiving care in this area)
* Age: 6 - 11 years
* Score > 1 standard deviation on the BHK deterioration score

Exclusion Criteria:

* Contraindication to the use of the tablet or virtual reality
* Moderate, severe or profound intellectual disability (Total Intelligence Quotient below 55 on an intellectual efficiency scale such as WISC-V or K-ABC-II).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-02-24 (Estimated); Study Completion 2027-02-24 (Estimated)

PRIMARY OUTCOMES:
Composite score brings together a set of parameters defining writing efficiency (static, kinematic and pressure) : Kaligo + | This assessment will be carried out twice a week up to 19 weeks during the baseline and intervention and once a week up to 1 month after the interventiona
  Static parameters: density, height, width and length Kinematic parameters: Time (in air and on paper), speed, number of speed inversion, median frequency of the speed, jerk and acceleration.
  Pressure: Median, 60th percentile, median frequency of the pressure change. The score is normalized between 0 (worst) and 1 (best).

SECONDARY OUTCOMES:
Assessing the ecological impact and its generalisation | This assessment will be conducted during the first week of the baseline, in the 10th week of the intervention, and once more one month after the intervention.
  Movement Assessment Battery for Children | Second Edition (M-ABC-II). Questionnaire to assess motor skills in everyday situations, comprising 3 parts: part A "movement in a static and/or predictable environment", part B "movement in a dynamic and/or non-static environment", part C "non-motor factors that can affect movement". A raw score is obtained for each of these parts, as well as a total motricity score (A + B).
Assessing the ecological impact and its generalisation | This assessment will be conducted during the first week of the baseline, in the 10th week of the intervention, and once more one month after the intervention
  Handwriting Proficiency Screening Questionnaire for Children (HPSQ-C). Questionnaire to assess motor skills in everyday situations, comprising 3 parts: part A "movement in a static and/or predictable environment", part B "movement in a dynamic and/or non-static environment", part C "non-motor factors that can affect movement". A raw score is obtained for each of these parts, as well as a total motricity score (A + B).
Assessing the ecological impact and its generalisation | This assessment will be conducted during the first week of the baseline, in the 10th week of the intervention, and once more one month after the intervention.
  Concise Assessment Scale for Children's Handwriting (BHK). In the BHK [Brave Handwriting Kindergarten], the child is asked to copy a text for 5 minutes. Blind double scoring is used (the scorer does not know when the child has copied the text). A degradation score is calculated: the higher the score, the more "degraded" the quality of the child's handwriting. The standardized score is taken into account for inclusion (to situate the child's performance in relation to his class), while the raw score is taken into account over the course of the intervention (allowing comparison of the subject with himself). Psychometric qualities are documented in the test manual.
Assessing the ecological impact and its generalisation | This assessment will be conducted during the first week of the baseline, in the 10th week of the intervention, and once more one month after the intervention.
  NEPSY-II is the only single measure that allows clinicians to create tailored assessments across six domains, specific to a child's situation SUBTESTS - ORIENTATION SUBTEST - VISUO-MOTOR PRECISION SUBTEST - INHIBITION SUBTEST - FACE RECOGNITION
Assessing the ecological impact and its generalisation | This assessment will be conducted during the first week of the baseline, in the 10th week of the intervention, and once more one month after the intervention.
  Purdue Pegboard Test (PPT). Test of manual dexterity and bimanual coordination. The child must place rods in holes on a board as quickly as possible, using the dominant hand, the non-dominant hand, then both hands simultaneously. In a final condition ("assembly"), the child must place a rod in one of the holes, then a washer, a tube and another washer, using both hands alternately. Raw scores (number of correctly placed and assembled pieces) are taken into account.
Assessing the ecological impact and its generalisation | This assessment will be conducted during the first week of the baseline, in the 10th week of the intervention, and once more one month after the intervention.
  Written Language Analytical Battery (BALE). In the BALE [Batterie Analytique du Langage Ecrit, Analytic test of the written language], the child is asked to write (under dictation) simple, complex and frequent irregular words from the French language, and to read regular and frequent irregular words. For the purposes of this study, only raw scores will be taken into account, in order to compare the subject with himself.
- Evaluate the maintenance of performance over time after the end of the intervention | This assessment will be carried out at the end of the intervention and every week for a month.
  Evolution of the Kaligo + score. Kaligo + Score: This composite score brings together a set of parameters defining writing efficiency (static, kinematic and pressure).
Assessing the specific nature of the intervention | This assessment will be conducted during the first week of the baseline, in the 10th week of the intervention, and once more one month after the intervention
  Evolution of performance on an untrained task. It will be demonstrated by the absence of as great an improvement in the control variable (face recognition task) compared with the improvement recorded in the primary endpoint
Assessing satisfaction with the intervention for the child and his or her family | during the last visit, 1 month after intervention
  The CSQ 8 is a short customer satisfaction questionnaire. The CSQ8 is the benchmark questionnaire for assessing satisfaction among parents, children and teenagers.
Assessing satisfaction with the intervention for the child and his or her family | during the last visit, 1 month after intervention
  10-point visual analogue scale to be completed by the child.
Assessing the acceptability and usability of the solution for families and professionals | during the last visit, 1 month after intervention
  Mobile Application Rating Scale (MARS). This validated questionnaire makes it possible to assess the quality of mobile healthcare applications in a way that is transparent for healthcare professionals and patients alike.
Assessing the acceptability and usability of the solution for families and professionals | during the last visit, 1 month after intervention
  System Usability Scale (SUS). This questionnaire is currently the most widely used in the scientific community for measuring user satisfaction with a product, interactive system or service.
Assessing the acceptability and usability of the solution for families and professionals | during the last visit, , 1 month after intervention
  Carrying out qualitative interviews with families and professionals

CONTACTS AND LOCATIONS:
Overall Officials: Christelle PONS BECMEUR, MP/PhD, Principal Investigator — Fondation Ildys
Locations (1):
- Fondation ILDYS, Brest, France

IPD SHARING:
Plan to Share IPD: No